CLINICAL TRIAL: NCT01983176
Title: Retrospective Clinical Outcome of Parotid Tumor Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201307054RIND
Record Dates: First submitted 2013-10-27; First posted 2013-11-13 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Parotid Tumors; Postoperative Complications
Keywords: Parotid tumor; Partial superficial parotidectomy; Facial palsy
MeSH Terms: conditions — Parotid Neoplasms; Postoperative Complications; Facial Paralysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to determine the histopathological results of parotid tumors and postoperative complications after partial superficial or total parotidectomy with facial nerve dissection and superficial musculoaponeurotic system reconstruction.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of parotid tumor
* Patients received the surgery of parotid tumor at NTUH by single surgeon ( Prof. Lou) from 2004/01 to 2012/12

Exclusion criteria:

-Inflammation or infection disease of parotid gland

Ages: 10 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent parotid surgery by a single operator in National Taiwan University Hospital from January 2004 to December 2012 were assessed for histopathological results and postoperative complications.
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Facial palsy | 6 months
  Record the grade of facial palsy in patients receiving the surgery of parotid tumor

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, MD, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan